CLINICAL TRIAL: NCT04208620
Title: A Phase 1 Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Cotadutide in Japanese Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Tolerability Study of Cotadutide in Japanese Obese Subjects With Type 2 Diabetes Melitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5671C00003
Record Dates: First submitted 2019-12-01; First posted 2019-12-23 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Cotadutide; MEDI0382; D5671C00003; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo
- Cotadutide (Experimental): Cotadutide administered subcutaneously
  Interventions: Drug: Cotadutide

INTERVENTIONS:
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo
Drug: Cotadutide — Cotadutide administered subcutaneously
  Arms: Cotadutide

SUMMARY:
This is a Phase 1 study designed to assess the safety and tolerability of MEDI0382 (Cotadutide) in Japanese T2DM patients.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study designed to evaluate the safety, tolerability, PK and efficacy of ascending doses of Cotadutide in Japanese obese subjects with T2DM. Approximately 20 subjects will be screened in total and 16 subjects will be randomized to Cotadutide or placebo in a 3:1 ratio. Those subjects who receive Cotadutide will be titrated up to HCTD. The study has a 2-week screening period, a run-in period of 9 days and an up to 7-week up-titration treatment period followed by a 3-week treatment extension period (if applicable), followed by a 28-day follow-up period.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated written informed consent prior to any mandatory study specific procedures, sampling, and analyses.
2. Subject must be 20 to 74 years of age at screening.
3. HbA1c range of 6.5% to 8.5% at screening and run-in visit.
4. Willing and able to self-inject investigational product for the duration of the study.
5. Individuals who are diagnosed with T2DM and have inadequate glycaemic control with diet and exercise.
6. Individuals whose current condition at enrolment are drug naïve defined as

   * Never received medical treatment for diabetes (insulin and/or other anti-diabetic agents [oral or injection]) OR
   * Received medical treatment for diabetes for less than 30 days since diagnosis.Subjects also should not have a history of insulin therapy within 2 weeks of screening (with the exception of insulin therapy during a hospitalization for other causes or use in gestational diabetes) OR
   * Previously received medical treatment for diabetes but have not been treated within 6 weeks of randomization.
7. BMI within the range 25 to 35 kg/m2 at screening.
8. Negative pregnancy test for female subjects.
9. Female subjects of childbearing potential who are sexually active with a male partner must be willing to use at least one highly effective method of contraception from screening and up to 4 weeks after the last dose of investigational product.

Exclusion Criteria

1. Subjects with any of the following results at screening and run-in visit
2. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study and/or any subject unable or unwilling to follow study procedures.
3. Acute pancreatitis at screening or history of chronic pancreatitis or serum triglyceride levels > 11 mmol/L (1000 mg/dL) at screening.
4. Significant inflammatory bowel disease, gastroparesis or other severe disease or surgery affecting the upper GI tract (including weight-reducing surgery and procedures), which may affect gastric emptying or could affect the interpretation of safety and tolerability data.
5. Significant hepatic disease (except for NASH or non-alcoholic fatty liver disease without portal hypertension or cirrhosis) and/or subjects with any of the following results at screening or run-in visit.

   * Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN)
   * Alanine transaminase (ALT) ≥ 3 × ULN
   * Total bilirubin (TBL) ≥ 2 × ULN
6. Impaired renal function defined as estimated glomerular filtration rate (GFR) < 60 mL/minute/1.73m2 at screening or run-in visit (GFR estimated according to Modification of Diet in Renal Disease [MDRD] using MDRD Study Equation IDMS-traceable [International System of Units (SI)]).
7. Poorly controlled hypertension defined as, For age ≤ 55 years; Systolic BP > 140 mmHg Diastolic BP ≥ 90 mmHg For age > 55 years; Systolic BP > 150 mmHg Diastolic BP ≥ 90 mmHg After 10 minutes of supine rest and confirmed by repeated measurement at screening or run-in visit. Subjects who fail BP screening criteria may be considered for 24-hour or day time ABPM at the discretion of the investigator. Subjects who maintain a mean 24-hour BP < 130/80 mmHg with a preserved nocturnal dip of > 15% or day time BP < 135/85 mmHg will be considered eligible
8. Resting heart rate is ≥ 80 bpm at screening or run-in visit.
9. Any clinically important abnormalities in rhythm, conduction, or morphology of the 12-lead ECG or any abnormalities that may interfere with the interpretation of serial ECG changes, including QTc interval changes at screening, as judged by the investigator.
10. Prolonged QT intervals corrected for heart rate using Fridericia's formula (QTcF) > 450 msec, or family history of long QT-segment at screening or run-in visit.
11. PR (PQ) interval prolongation (> 220 msec), intermittent second (Wenckebach block while asleep is not exclusive), or third-degree atrioventricular (AV) block, or AV dissociation at screening or run-in visit.
12. Persistent or intermittent complete bundle branch block. A QRS duration < 120 msec is acceptable if there is no evidence of ventricular hypertrophy or preexcitation at screening or run-in visit.
13. Abnormal findings during the exercise stress test, such as chest pain, dyspnoea, presyncope, arrhytmias, signs of cardiac ischemia on ECG as judged by the investigator.
14. History of, unstable angina pectoris, myocardial infarction, transient ischemic attack, or stroke, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft or who are due to undergo these procedures at the time of screening.
15. Severe congestive heart failure (New York Heart Association Class III or IV).
16. Basal calcitonin level > 50 ng/L at screening, or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia.
17. Hemoglobinopathy, hemolytic anemia or chronic anemia (hemoglobin, < 11.5 g/dL [115 g/L]) for males, < 10.5 g/dL (105 g/L) for females) at screening or run-in visit, or any other condition known to interfere with the interpretation of HbA1c measurement.
18. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer.
19. Any positive results for serum hepatitis B surface antigen, hepatitis C antibody, and human HIV antibody.
20. History of substance dependence, alcohol abuse, or excessive alcohol intake (defined as an average weekly intake of > 21 alcoholic drinks for men or > 10 alcoholic drinks for women) within 3 years prior to screening and/or a positive screen for drugs of abuse or alcohol at screening or run-in visit. Subjects who use benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
21. Symptoms of depression or any other psychiatric disorder requiring treatment with medication (eg, anti-depressants, anti-psychotics) at screening. However, subjects who use benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
22. History of severe allergy/hypersensitivity, including to any component of the investigational product formulation including excipients or other biological agent, any of the proposed study treatments, or ongoing clinically important allergy/hypersensitivity.
23. Any subject who has received another investigational product as part of a clinical study or a GLP-1 analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening.
24. Any subject who has received any of the following medications within the specified timeframe prior to the start of the study.

    * Herbal preparations within one week prior to the start of screening or drugs licensed for control of body weight or appetite within 30 days (or 5 half-lives of the drug) prior to the start of screening
    * Opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying and within 2 weeks prior to the start of dosing
    * Antimicrobials within the quinolone, macrolide or azole class within 2 weeks prior to the start of dosing
    * Any change in antihypertensive medication within 3 months prior to screening
    * Any change in thyroid replacement therapy within 2 months prior to screening
    * Aspirin at a total daily dose of greater than 150 mg
    * Paracetamol or paracetamol-containing preparations at a total daily dose of greater than 3000 mg
    * Ascorbic acid (vitamin C) supplements at a total daily dose of greater than 1000 mg
25. Concurrent participation in another study of any kind and repeat randomization in this study.
26. Received Cotadutide in another clinical study prior to enrolment in this study.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Incidence of treatment-emergent serious adverse events (TESAEs) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Clinically important changes in 12-lead electrocardiogram (ECG) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Vital signs as measured by pulse rate (bpm) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Vital signs as measured by blood pressure (mmHg) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
ABPM (Ambulatory blood pressure monitoring) to measure pulse rate (bpm) and blood pressure (mmHg) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Physical examination (abnormality to be reported as part of adverse events) | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide
Clinical laboratory evaluations | Baseline until the follow-up period, 28 days post-last dose
  To assess the safety and tolerability of Cotadutide

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) during the dosing interval (AUCtau) | Day1 of Up-titration treatment period to Day 21 of Treatment extension period, total of up to 10 weeks
  To characterize the PK profile of Cotadutide
Maximum observed concentration (Cmax) | Day1 of Up-titration treatment period to Day 21 of Treatment extension period, total of up to 10 weeks
  To characterize the PK profile of Cotadutide
Time to Cmax (tmax) | Day1 of Up-titration treatment period to Day 21 of Treatment extension period, total of up to 10 weeks
  To characterize the PK profile of Cotadutide
Trough plasma concentration (Ctrough) | Day1 of Up-titration treatment period to Day 21 of Treatment extension period, total of up to 10 weeks
  To characterize the PK profile of Cotadutide
Anti-drug antibodies (ADAs) to Cotadutide | At baseline through end of study, 98 days in total
  To characterize the immunogenicity of Cotadutide
Change in average glucose levels (mg/dL) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in coefficient of variation | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in hyperglycemia (> 140 mg/dL) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in normoglycemia (70 -140 mg/dL) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in clinically significant hypoglycemia (< 54 mg/dL) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in estimated hemoglobin A1c (HbA1c) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in fasting plasma glucose (mg/dL) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by additional measrues of glucose control
Change in HbA1c | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on glucose control as measured by additional measrues of glucose control
Percentage change in body weight | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on body weight
Absolute change in body weight (kg) | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on body weight
Proportion of subjects achieving > 5% body weight loss | At baseline through end of study, 98 days in total
  To assess the effect of Cotadutide on body weight

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home